CLINICAL TRIAL: NCT05226650
Title: The Effect of Irregular Meal Pattern on Nitrogen Balance: a Randomized Controlled Trial in Healthy Normal-weight Women
Brief Title: The Effect of Irregular Meal Pattern on Nitrogen Balance in Healthy Normal-weight Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Moira Taylor, Dr Moira A Taylor, University of Nottingham
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 189-1812
Record Dates: First submitted 2021-02-19; First posted 2022-02-07 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Nitrogen Balance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Regular meal pattern (Experimental): Participants will follow a regular meal pattern for a week
  Interventions: Other: Regular meal pattern
- Irregular meal pattern (Experimental): Participants will follow an irregular meal pattern for a week
  Interventions: Other: Irregular meal pattern

INTERVENTIONS:
Other: Regular meal pattern — 6 meals every day
  Arms: Regular meal pattern
Other: Irregular meal pattern — It consists of consuming a different number of meals every day (between 3 and 9).
  Arms: Irregular meal pattern

SUMMARY:
Nitrogen balance (NB) is defined as the net difference between the intake of nitrogen (input) and its excretion (output). NB was considered as an indicator of the catabolic stress level. Thus, a negative NB can occur as a result of catabolism which leads to muscle mass loss. It was demonstrated that there is a relationship between meal frequency and N loss. Irregular meal patterns have been considered as a possible new risk factor for obesity and its consequences, specifically cardiovascular disease and metabolic syndromes. As the regular meal pattern is associated with higher BMI in many observational studies and has an impact on the metabolism of carbohydrates and lipids, it could also affect protein metabolism.

Eating irregularly can cause chrono-disruption because the changes in the timing of food intake as a consequence may also alter the chrono-biological or circadian rhythm of many hormones such as insulin, glucagon, adiponectin, leptin and gastric acid secretion. From this, investigators hypothesized that following an irregular meal pattern can negatively influence the N balance and circadian rhythm.

DETAILED DESCRIPTION:
The study will have a crossover randomised, non blinded two meal pattern design with healthy adult female volunteers recruited from Nottingham, UK and the surrounding area.

Firstly, a screening visit lasting approximately an hour will be arranged and height, weight, and waist circumference will be measured following standard procedures (eg without shoes, wearing light clothes). Body composition will be obtained using skinfold thickness at four sites (triceps, biceps, subscapular and suprailiac). A blood sample (8 ml) will be obtained for routine blood investigation. A number of questionnaires will be completed to assess medical health, sleep duration, physical activity levels, eating behaviour and depression. On departure, subjects will be asked to complete a 4 days food diary.

The present study will last for 5 weeks. During the first week participants will be required to adopt one of two meal patterns, followed by a three week washout period, in which they will be allowed to return to their habitual diet, before undertaking a second week intervention following the second meal pattern. These meal patterns will consist of consuming 1) a regular meal pattern of 6 daily meals for two weeks, or 2) an irregular one consisting of consuming a different number of meals every day (between 3 and 9). Investigators propose to provide an iso-energetic diet containing identical foods with macronutrient composition (as a percentage of total energy per day) of 50% carbohydrate, 35% fat, and 15% protein for both patterns. All foods to be consumed during the study (1st and 5th week) will be provided free of charge. These will comprise foods commonly consumed in the British diet and will be consumed in amounts designed to keep body weight constant during the study. Participants will complete a food compliance diary over the study period. Physical activity will be captured by BodyMedia SenseWear armband to ensure that participants have a similar physical activity level in both intervention periods. This device records and analyses physiological parameters, and uses algorithms to report daily movement, calories burned, degree of physical activity and steps taken. It will be placed on the back of the upper left arm (the tricep). The Armband logo must face upward towards the shoulder and the silver sensors on the underside of the Armband will be in contact with skin.

Participants will be advised to consume a standardized evening meal based on their food record on the day before the start of each intervention and to provide 7, 24-h urine samples over the course of each intervention period. All urine was collected from study participants for 24 hr beginning at 7 am. Urine will be collected into 7 plastic urine containers without preservative. 5 ml will be stored from the well-mixed 24-h urine collection and analysed for urinary urea. In addition, they will be advised to wear a wireless iButton data logger to measure the wrist temperature in order to assess the circadian rhythm. The iButtons will be programmed to sample every 10 min, and will be attached to a double-sided cotton sport wrist band usingVelcro®, with the sensor face of the iButton being placed over the inside of the wrist, on the radial artery of the non-dominant hand.

Finally, subjective appetite (including hunger, fullness and desire to eat) will be assessed using visual analogue scales (VAS) during the intervention. Participants will be provided with a booklet in which to record the subjective appetite before and after each single meal on day 7 during both intervention periods when the subjects consume 6 meals/d during each intervention.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5 and 25 kg/m2,
* Age between 18 and 40y,
* Non-smokers,
* Non high-alcohol consumers (≥ 14 units/week),
* Regular menstruation or on the oral contraceptive pills,
* Their weight is stable during the previous 3 months,
* No self-reported history of serious medical conditions and not under medication.

Exclusion Criteria:

* Pregnant or lactating women
* Smokers
* High-alcohol consumers (≥ 14 units/week)
* Subjects with high score for depression using Becks Depression Inventory
* subjects Eating Attitudes Test (EAT-26) score >20
* Subjects who on diet or seeking to lose weight
* Subjects with high consumption of coffee or tea > 3 cups/day

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2019-09-13 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Nitrogen balance | 7 days
  Nitrogen balance will be calculated using urinary urea nitrogen which will be estimated from 24 hour urinary urea excretion

SECONDARY OUTCOMES:
Subjective appetite | Before and after each single meal on day 7 during both intervention periods
  It (including hunger, fullness and desire to eat) will be assessed during the intervention using a 100 mm scale. 100 mm represents the highest experience possible of the sensation and 0 represents no experience of the sensation. Participants were provided with a booklet in which to record the subjective appetite before and after each single meal on day 7 during both intervention periods when the subjects consume 6 meals/d during each intervention
Wrist temperature | 7 days
  Wrist temperature will be assessed using a wireless wrist iButton

CONTACTS AND LOCATIONS:
Overall Officials: Ian Macdonald, PhD, Study Director — University of Nottingham
Locations (1):
- The University of Nottingham, Nottingham, County (optional), United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymised individual personal data will be shared, upon specific request from other researchers, for example, in order to undertake a meta analysis
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: when requested
Access Criteria: On receipt of requests, data will be made accessible if agreed by the University of Nottingham

REFERENCES:
- [Background] Alhussain MH, Macdonald IA, Taylor MA. Irregular meal-pattern effects on energy expenditure, metabolism, and appetite regulation: a randomized controlled trial in healthy normal-weight women. Am J Clin Nutr. 2016 Jul;104(1):21-32. doi: 10.3945/ajcn.115.125401. Epub 2016 Jun 15. PMID 27305952
- [Background] Dickerson, R. N. (2005). Using nitrogen balance in clinical practice. Hospital Pharmacy, 40(12), 1081-1087
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Regular meal frequency creates more appropriate insulin sensitivity and lipid profiles compared with irregular meal frequency in healthy lean women. Eur J Clin Nutr. 2004 Jul;58(7):1071-7. doi: 10.1038/sj.ejcn.1601935. PMID 15220950
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Decreased thermic effect of food after an irregular compared with a regular meal pattern in healthy lean women. Int J Obes Relat Metab Disord. 2004 May;28(5):653-60. doi: 10.1038/sj.ijo.0802616. PMID 15085170
- [Background] Farshchi HR, Taylor MA, Macdonald IA. Beneficial metabolic effects of regular meal frequency on dietary thermogenesis, insulin sensitivity, and fasting lipid profiles in healthy obese women. Am J Clin Nutr. 2005 Jan;81(1):16-24. doi: 10.1093/ajcn/81.1.16. PMID 15640455
- [Background] Garrow JS, Durrant M, Blaza S, Wilkins D, Royston P, Sunkin S. The effect of meal frequency and protein concentration on the composition of the weight lost by obese subjects. Br J Nutr. 1981 Jan;45(1):5-15. doi: 10.1079/bjn19810072. PMID 7470437
- [Background] McGinnis GR, Young ME. Circadian regulation of metabolic homeostasis: causes and consequences. Nat Sci Sleep. 2016 May 27;8:163-80. doi: 10.2147/NSS.S78946. eCollection 2016. PMID 27313482
- [Background] Pot GK, Hardy R, Stephen AM. Irregular consumption of energy intake in meals is associated with a higher cardiometabolic risk in adults of a British birth cohort. Int J Obes (Lond). 2014 Dec;38(12):1518-24. doi: 10.1038/ijo.2014.51. Epub 2014 Mar 28. PMID 24675713
- [Background] Pot GK, Hardy R, Stephen AM. Irregularity of energy intake at meals: prospective associations with the metabolic syndrome in adults of the 1946 British birth cohort. Br J Nutr. 2016 Jan 28;115(2):315-23. doi: 10.1017/S0007114515004407. Epub 2015 Nov 9. PMID 26548599